CLINICAL TRIAL: NCT04852510
Title: Amelioration of Polycystic Ovary Syndrome Related Disorders by Supplementation of Thymoquinone and Metformin
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Saudi German Hospital - Madinah (Other)
Responsible Party: Principal Investigator, Islam Mohamed Magdi Ammar, Associate Professor and Consultant of Obstetrics and Gynecology, Saudi German Hospital - Madinah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGHM-JAN2019-OBGYN
Record Dates: First submitted 2021-04-09; First posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — thymoquinone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Metformin 500 mg three times daily (5) with meals for 6 months (Metfor® 500 mg, Metformin hydrochloride tablets. TABUK Pharmaceutical. KSA).
  Interventions: Drug: Metformin Versus a combination of Metformin and Thymoquinone (TQ)
- Group B (Active Comparator): A combination of Metformin 500 mg three times daily with meals (Metfor® 500 mg, Metformin hydrochloride tablets. TABUK Pharmaceutical. KSA) and Thymoquinone (TQ) in the form of Black Cumin oil (Cumin Mar® Black cumin oil 500 mg soft gel capsules, MARNYS. Spain) three times daily before meals for 6 months.
  Interventions: Drug: Metformin Versus a combination of Metformin and Thymoquinone (TQ)

INTERVENTIONS:
Drug: Metformin Versus a combination of Metformin and Thymoquinone (TQ) — Patients were divided into two groups (A and B) using a computer-based software Open Epi version 3.21. Patients in Group A, received Metformin 500 mg three times daily (5) with meals for 6 months (Metfor® 500 mg, Metformin hydrochloride tablets. TABUK Pharmaceutical. KSA). Patients in Group B, received a combination of Metformin 500 mg three times daily with meals (Metfor® 500 mg, Metformin hydrochloride tablets. TABUK Pharmaceutical. KSA) and Thymoquinone (TQ) in the form of Black Cumin oil (Cumin Mar® Black cumin oil 500 mg soft gel capsules, MARNYS. Spain) three times daily before meals for 6 months.
  Other Names: Metfor® 500 mg, Metformin hydrochloride tablets. TABUK Pharmaceutical. KSA; Cumin Mar® Black cumin oil 500 mg soft gel capsules, MARNYS. Spain

SUMMARY:
Objective: To investigate the potential benefit of adding Thymoquinone to Metformin in alleviating symptoms of polycystic ovarian syndrome.

Methods: 207 overweight and obese PCOS Patients were divided into two groups. Patients in Group A, received Metformin 500 mg three times daily for 6 months. Patients in Group B, received a combination of Metformin 500 mg and Thymoquinone in the form of Black Cumin oil 500 mg capsules three times daily for 6 months. Follow up was done after 3 and 6 months from the beginning of the study for evaluation of menstrual cycle pattern, body mass index, Waist circumference, Hip circumference, and Waist / Hip ratio, Oral glucose tolerance test, Glycosylated Hemoglobin A1C, Superoxide dismutase activity and Malondialdehyde concentration.

DETAILED DESCRIPTION:
This randomized clinical trial was conducted in the department of Obstetrics and Gynaecology at the Saudi German Hospital, Madinah-KSA, during the period from February 2019 to August 2020. The study included 207 patients who fulfilled the following inclusion criteria: age of 18 to 35 years, overweight and obese PCOS patients (overweight defined as body mass index (BMI) 25-29.9 kg/m2 and obesity defined as BMI ≥ 30 kg/m2) attending the outpatient clinic, complaining of amenorrhea or oligomenorrhea with or without hirsutism. Amenorrhea was defined as absence of menstruation for six or more months. Oligomenorrhea was defined as cycle interval of more than 35 days but less than 6 months. PCOS was diagnosed according to the 2004 Rotterdam ESHRE/ASRM Consensus workshop, with presence of at least 2 out of 3 criteria: oligo- and/or anovulation, clinical and/or biochemical hyperandrogenism, and polycystic ovarian morphology identified by ultrasound with more than 12 small antral follicles in an ovary, with exclusion of other related aetiologies like androgen-secreting tumours, congenital adrenal hyperplasia, and hyperprolactinemia. Prediabetes patients who are at increased risk of developing diabetes, as defined by the American Diabetes Association 2014, were included. Those patients had; impaired fasting glucose (IFG) defined as fasting plasma glucose (FPG) levels of 100 to 125 mg/dL (Fasting was described as no caloric intake for at least 8 hours), or impaired glucose tolerance (IGT) defined as 2-hour readings of 140 to 199 mg/dL in the oral glucose tolerance test (OGTT). Patients who were considered at very high risk of developing diabetes according to the International Expert Committee 2009 were also included. Those patients had their Glycosylated Hemoglobin A1C levels between 5.7% and 6.4%.

Exclusion criteria were: lean or average weight PCOS with BMI < 25 kg/m2, morbidly obese patients with BMI ≥ 35 kg/m2, patients suffering from any other metabolic disorders, history of receiving any hormonal treatment or any drug affecting carbohydrate metabolism 3 months prior to the beginning of the study, and inability to attend the regular follow up visits. Already known and recently diagnosed diabetic patients were excluded from the study. According to the American Diabetes Association 2014, diabetes mellitus was defined as Glycosylated Hemoglobin A1C levels ≥ 6.5% or FPG ≥ 126 mg/dL or 2-hour plasma glucose readings ≥ 200 mg/dL during 75 g OGTT, or presence of classic symptoms of hyperglycemia with random plasma glucose levels ≥ 200 mg/dL. Thyroid diseases and hyperprolactinemia were treated before participation.

The Study was in accordance with the Helsinki declaration 1964 and its later amendments. The study protocol was approved by the local ethics committee. All patients signed an informed consent before participation.

During the first booking visit, initial assessment was carried out with detailed history taking, including personal, medical, surgical, obstetric and menstrual history. General examination was done with measurement of BMI, waist circumference (WC), hip circumference (HC) and waist: hip ratio (WHR).

BMI had the disadvantage of not truly representing the body fat distribution and hence the nature of obesity as concluded by many studies. So, the waist circumference, hip circumference and waist: hip ratio were selected as more convenient measures of abdominal visceral fat and hence important clinical markers to predict patients at risk of developing DM and cardiovascular diseases.

Measurements were carried out according to the World Health Organization (WHO) STEPS protocol 2008. Waist circumference was measured at the midpoint between the lower margin of the last palpable rib and the top of the iliac crest. Hip circumference was measured around the widest portion of the buttocks. For both measurements, the tape was adjusted parallel to the floor at the level at which the measurement was made. The tape was held snugly around the body, but not pulled so tight. The patient was standing with feet close together, arms at the sides and body weight evenly distributed across the feet. The waist circumference was measured at the end of a normal expiration, when the lungs are at their functional residual capacity. Because many individuals unconsciously react to waist measurements by sucking their abdominal wall, the patients were advised to relax and take a few natural breaths before the actual measurement was made. Each measurement was repeated twice; if the measurements were within 1 cm of one another, the average was calculated. If the difference between the two measurements exceeded 1 cm, the two measurements were repeated.

During the booking visit; a basal pelvic ultrasound was done for virgin participants and transvaginal ultrasound (TVS) for non-virgin patients. Blood samples were also collected for OGTT, Glycosylated Hemoglobin A1C levels, estimation of SOD activity and MDA concentrations.

The oral glucose tolerance test (OGTT) was performed in the morning after an overnight fasting of at least 8 hours, utilizing a glucose load containing the equivalent of 75 grams of anhydrous glucose dissolved in water. Glycosylated Hemoglobin A1C levels were also measured.

For estimation of SOD activity, centrifugation of the blood samples was done at 1000 g for 10 minutes, the serum was frozen and stored at -80 °C until the time of analysis. SOD activity was based on the ability of the enzyme to inhibit the reduction of nitro blue tetrazolium dye mediated by phenazine methosulphate. The purified SOD inhibits the initial rate of reduction of (O2 to O2-) mediated by the activated phenazine methosulphate which then reduces the nitro blue tetrazolium. The percentage of inhibition was then calculated and compared to the standard of 0.5 μg of the enzyme that produced inhibition of 80 % (activity = 3.000 units/mg protein). The SOD activity was finally expressed as units of enzymatic activity per mg of protein contained in the samples (U/mg protein).

Malondialdehyde (MDA) concentrations were measured in µmol/liter using the derivatization MDA with thiobarbituric acid (TBA) based on spectrophotometric determination of pink fluorescent MDA-TBA complex produced after reaction with 2-thiobarbituric acid at high temperature and low pH. The assay kits for MDA and SOD were products of (Cell Biolabs Inc, San Diego, USA).

Patients were divided into two groups (A and B) using a computer-based software Open Epi version 3.21. Patients in Group A, received Metformin 500 mg three times daily (5) with meals for 6 months (Metfor® 500 mg, Metformin hydrochloride tablets. TABUK Pharmaceutical. KSA). Patients in Group B, received a combination of Metformin 500 mg three times daily with meals (Metfor® 500 mg, Metformin hydrochloride tablets. TABUK Pharmaceutical. KSA) and Thymoquinone (TQ) in the form of Black Cumin oil (Cumin Mar® Black cumin oil 500 mg soft gel capsules, MARNYS. Spain) three times daily before meals for 6 months.

Patients were instructed not to receive any non-study drug during the study period, to increase their physical activity by performing aerobic physical exercise (moderate level for two hours and thirty minutes weekly or vigorous level for one hour and fifteen minutes weekly) divided over at least three days of the week, and to consume a low caloric diet.

All patients were advised to attend for follow up after 3 and 6 months from the beginning of the study for evaluation of their BMI, waist circumference, hip circumference, and waist / hip ratio and to withdraw a blood sample for OGTT, A1C, SOD activity and MDA concentration. Patients were also asked about their menstrual cycle pattern.

The primary study outcomes were; the resumption of regular menstrual cycles, weight reduction as detected by decreased BMI, change of body fat distribution as proved by reduced Waist/Hip ratio, improvement of the glycemic control as documented by normalization of OGTT and A1C and regaining the normal oxidative balance as evidenced by decreased MDA concentration and increased SOD activity.

ELIGIBILITY:
Inclusion criteria:

* Age of 18 to 35 years
* Overweight and obese PCOS patients (overweight defined as body mass index (BMI) 25-29.9 kg/m2 and obesity defined as BMI ≥ 30 kg/m2).
* History of amenorrhea or oligomenorrhea with or without hirsutism. Amenorrhea was defined as absence of menstruation for six or more months. Oligomenorrhea was defined as cycle interval of more than 35 days but less than 6 months.
* PCOS diagnosed according to the 2004 Rotterdam ESHRE/ASRM Consensus workshop, with presence of at least 2 out of 3 criteria: oligo- and/or anovulation, clinical and/or biochemical hyperandrogenism, and polycystic ovarian morphology identified by ultrasound with more than 12 small antral follicles in an ovary.
* Prediabetes defined by the American Diabetes Association 2014, as fasting plasma glucose (FPG) levels of 100 to 125 mg/, or impaired glucose tolerance (IGT) defined as 2-hour readings of 140 to 199 mg/dL in the oral glucose tolerance test (OGTT). Also, patients who had their Glycosylated Hemoglobin A1C levels between 5.7% and 6.4%.

Exclusion criteria were:

* Lean or average weight PCOS with BMI < 25 kg/m2, morbidly obese patients with BMI ≥ 35 kg/m2.
* Patients suffering from any other metabolic disorders.
* History of receiving any hormonal treatment or any drug affecting carbohydrate metabolism 3 months prior to the beginning of the study.
* Inability to attend the regular follow up visits.
* Already known and recently diagnosed diabetic patients. According to the American Diabetes Association 2014 (16), diabetes mellitus was defined as Glycosylated Hemoglobin A1C levels ≥ 6.5% or FPG ≥ 126 mg/dL or 2-hour plasma glucose readings ≥ 200 mg/dL during 75 g OGTT, or presence of classic symptoms of hyperglycemia with random plasma glucose levels ≥ 200 mg/dL.
* Thyroid diseases
* Hyperprolactinemia

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 253 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
The change of menstrual cycle pattern. | At the beginning of the study, After 3 months and After 6 Months
  Patients were asked about their menstrual cycle pattern (Frequency of menstrual cycles and number of days of menses). Resumption of normal menstrual cyclicity was defined as having menses every 3-5 weeks. Amenorrhea was defined as absence of menstruation for six or more months. Oligomenorrhea was defined as cycle interval of more than 35 days but less than 6 months.
The change of body mass index (BMI). | At the beginning of the study, After 3 months and After 6 Months
  The body mass index is calculated as the body weight in kilograms divided by the height in meters squared. Normal BMI was defined as a range of 18.5-24.9 kg/m2. Overweight defined as body mass index (BMI) 25-29.9 kg/m2 and obesity defined as BMI ≥ 30 kg/m2.
Change of body fat distribution as proved by change of Waist/Hip ratio. | At the beginning of the study, After 3 months and After 6 Months
  Waist circumference was measured at the midpoint between the lower margin of the last palpable rib and the top of the iliac crest. Hip circumference was measured around the widest portion of the buttocks. For both measurements, the tape was adjusted parallel to the floor at the level at which the measurement was made. The tape was held snugly around the body, but not pulled so tight. The patient was standing with feet close together, arms at the sides and body weight evenly distributed across the feet. The waist circumference was measured at the end of a normal expiration, when the lungs are at their functional residual capacity. Each measurement was repeated twice; if the measurements were within 1 cm of one another, the average was calculated. If the difference between the two measurements exceeded 1 cm, the two measurements were repeated.
Change of oral glucose tolerance test (OGTT) results. | At the beginning of the study, After 3 months and After 6 Months
  The oral glucose tolerance test (OGTT) was performed in the morning after an overnight fasting of at least 8 hours, utilizing a glucose load containing the equivalent of 75 grams of anhydrous glucose dissolved in water. Prediabetes was defined by the American Diabetes Association 2014 as those patients who have; impaired fasting glucose (IFG) defined as fasting plasma glucose (FPG) levels of 100 to 125 mg/dL (Fasting was described as no caloric intake for at least 8 hours), or impaired glucose tolerance (IGT) defined as 2-hour readings of 140 to 199 mg/dL in the oral glucose tolerance test (OGTT). Diabetes mellitus was defined According to the American Diabetes Association 2014, as FPG ≥ 126 mg/dL or 2-hour plasma glucose readings ≥ 200 mg/dL during 75 g OGTT.
Change of Glycosylated Hemoglobin A1C levels. | At the beginning of the study, After 3 months and After 6 Months
  Glycosylated Hemoglobin A1C levels were measured as percentage (%) from the total hemoglobin. Normal range defined as readings below 5.7%. Prediabetes was defined by the American Diabetes Association 2014 as patients who have their Glycosylated Hemoglobin A1C levels between 5.7% and 6.4%. Diabetes mellitus was defined According to the American Diabetes Association 2014, as Glycosylated Hemoglobin A1C levels ≥ 6.5%.
Change of serum Malondialdehyde (MDA) concentrations. | At the beginning of the study, After 3 months and After 6 Months
  Malondialdehyde (MDA) concentrations were measured in µmol/liter using the derivatization MDA with thiobarbituric acid (TBA) based on spectrophotometric determination of pink fluorescent MDA-TBA complex produced after reaction with 2-thiobarbituric acid at high temperature and low pH. The assay kits for MDA and SOD were products of (Cell Biolabs Inc, San Diego, USA).
Change of serum superoxide dismutase (SOD) activity. | At the beginning of the study, After 3 months and After 6 Months
  For estimation of SOD activity, centrifugation of the blood samples was done at 1000 g for 10 minutes, the serum was frozen and stored at -80 °C until the time of analysis. SOD activity was based on the ability of the enzyme to inhibit the reduction of nitro blue tetrazolium dye mediated by phenazine methosulphate. The purified SOD inhibits the initial rate of reduction of (O2 to O2-) mediated by the activated phenazine methosulphate which then reduces the nitro blue tetrazolium. The percentage of inhibition was then calculated and compared to the standard of 0.5 μg of the enzyme that produced inhibition of 80 % (activity = 3.000 units/mg protein). The SOD activity was finally expressed as units of enzymatic activity per mg of protein contained in the samples (U/mg protein).

CONTACTS AND LOCATIONS:
Overall Officials: Islam Mohamed Magdi Ammar, M.D., Principal Investigator — Saudi German Hospital - Madinah
Locations (1):
- Saudi German Hospital, Al Madīnah, Madinah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No